CLINICAL TRIAL: NCT00467623
Title: Holotranscobalamin Remains Unchanged During Pregnancy. Longitudinal Changes of Cobalamins and Its Binding Proteins During Pregnancy and Postpartum
Brief Title: Holotranscobalamin Remains Unchanged During Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other)
Other Study IDs: KA-93140
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2007-04

CONDITIONS: Vitamin B12 Deficiency
Keywords: Pregnancy; holotranscobalamin; cobalamin; vitamin B12 analogues; reference interval
MeSH Terms: conditions — Vitamin B 12 Deficiency

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background and objective: Plasma cobalamins decrease during pregnancy but it is not fully elucidated how this is reflected in the total and cobalamin saturated transport proteins, transcobalamin (total TC, holoTC) and haptocorrin (total HC, holoHC). TC transports cobalamin into the cells. The function of HC is unknown, but in contrast to TC it binds both cobalamins and cobalamin analogues.

Design and methods: Healthy pregnant women (N=141) had blood samples drawn at 18th, 32nd, 39th gestation week and 8 weeks postpartum. The protein moiety of TC and HC (total and holo) was measured by in-house ELISA methods.

DETAILED DESCRIPTION:
Background and objective: Plasma cobalamins decrease during pregnancy but it is not fully elucidated how this is reflected in the total and cobalamin saturated transport proteins, transcobalamin (total TC, holoTC) and haptocorrin (total HC, holoHC). TC transports cobalamin into the cells. The function of HC is unknown, but in contrast to TC it binds both cobalamins and cobalamin analogues.

Design and methods: Healthy pregnant women (N=141) had blood samples drawn at 18th, 32nd, 39th gestation week and 8 weeks postpartum. The protein moiety of TC and HC (total and holo) was measured by in-house ELISA methods.

ELIGIBILITY:
Inclusion Criteria:

* Danish healthy Caucasian women >18 years of age with previous uncomplicated pregnancies and deliveries and presently with a normal pregnancy.

Exclusion Criteria:

* >4 cigarettes smoked per day,
* Treatment with vitamin B12, folic acid or acetyl salicylic acid,
* Impaired renal function and clinically significant vaginal haemorrhage before first visit as well as blood haemoglobin <6.4 mmol/L at first visit.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150
Dates: Start 1995-01; Study Completion 1997-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nils Milman, MD, Principal Investigator — University of Copenhagen
Locations (1):
- Nils Milman, Copenhagen, Denmark